#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for an open label parallel group study to investigate the optimum methodology for the use of LPS or GM-CSF as challenge agents on healthy participants by assessing inflammatory biomarkers in cantharidin-induced skin blisters, peripheral blood, and urine. |
| <b>Compound Number</b> | : | No Compound (Study 207654) |
| <b>Effective Date</b> | : | 14-MAY-2018 |

# **Description:**

- This version of the RAP is intended to describe the safety and biomarker analyses required for dose escalation and planned biomarker analyses required for interim analyses for study 207654. A subsequent version of the RAP will be developed for Final study reporting.
- Only sections related to dose escalation and interim analyses have been described.

#### **RAP Author(s):**

| Approver | Date | Approval Method |
|-------------------------------------------|------|-----------------|
| PPD | | |
| Senior Statistician | N/A | N/A |
| (Immuno-Inflammation Clinical Statistics) | | |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Associate Programmer (Immuno-Inflammation Clinical Programming) | 11-May-2018 | eTMF |
| VP Medicine Development Leader | 12-May-2018 | eTMF |
| Director, SERM | 11-May-2018 | eTMF |
| Principal Clinical Research Scientist (CPSSO) | 14-May-2018 | eTMF |
| Data Manager (CPSSO) | 11-May-2018 | eTMF |
| Director of Scientific Operations (CPSSO) | 11-May-2018 | e-Mail |
| Scientific Leader (Epigenetics DPU) | 11-May-2018 | e-Mail |
| Head of Medicinal Chemistry & Early Development Leader (MM DPU) | 13-May-2018 | e-Mail |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Statistical Leader (Immuno-Inflammation Clinical Statistics) | 11-May-2018 | eTMF |
| Biostatistics and Programming Manager (Immuno-Inflammation Clinical Programming) | 13-May-2018 | eTMF |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 5 |
| 2. | SUMN<br>2.1. | MARY OF KEY PROTOCOL INFORMATION | |
| | 2.2.<br>2.3. | Study Objective(s) and Endpoint(s) | 6 |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | | NED ANALYSES | |
| | 3.1.<br>3.2. | Dose Escalation | |
| | 3.2.<br>3.3. | Interim AnalysesFinal Analyses | |
| 4. | ANAL | YSIS POPULATIONS | 13 |
| | 4.1. | Protocol Deviations | 14 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING /ENTIONS | 15 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Examination of Covariates, Other Strata and Subgroups | |
| | 0.0. | 5.3.1. Covariates and Other Strata | |
| | | 5.3.2. Examination of Subgroups | |
| | 5.4. | Multiple Comparisons and Multiplicity | 16 |
| | 5.5. | Other Considerations for Data Analyses and Data Handling Conventions | 16 |
| 6. | STUD | Y POPULATION ANALYSES | 17 |
| 0. | 6.1. | Overview of Planned Study Population Analyses | |
| 7. | | CACY ANALYSES | |
| | 7.1. | Primary Biomarker Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | <ul><li>7.1.4. Strategy for Intercurrent (Post-Randomization) Events</li><li>7.1.5. Statistical Analyses / Methods</li></ul> | |
| | 7.2. | Secondary Biomarker Analyses | |
| | 1.2. | 7.2.1. Endpoint / Variables | |
| | | 7.2.2. Summary Measure | |
| | | 7.2.3. Population of Interest | |
| | | 7.2.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.2.5. Statistical Analyses / Methods | |
| | 7.3. | Exploratory Biomarker Analyses | 20 |
| 8. | SAFE | TY ANALYSES | 21 |
| 9. | RFFF | RENCES | 22 |


| 0. | APPEI | NDICES. | | 23 |
|---|---|---|---|---|
| | 10.1. | Appendi | x 1: Schedule of Activities | 23 |
| | | 10.1.1. | Protocol Defined Schedule of Events | 23 |
| | 10.2. | Appendi | x 2: Data Display Standards & Handling Conventions | <mark>24</mark> |
| | | 10.2.1. | Reporting Process | |
| | | 10.2.2. | Reporting Standards | <mark>24</mark> |
| | 10.3. | Appendi | x 3: Derived and Transformed Data | <mark>26</mark> |
| | | 10.3.1. | General | <mark>26</mark> |
| | | 10.3.2. | Study Population | 26 |
| | | 10.3.3. | Biomarker | 26 |
| | 10.4. | Appendi | x 4: Reporting Standards for Missing Data | 34 |
| | | 10.4.1. | Premature Withdrawals | 34 |
| | | 10.4.2. | Handling of Missing Data | 34 |
| | | | 10.4.2.1. Handling of Missing and Partial Dates | 34 |
| | 10.5. | Appendi | x 5: Values of Potential Clinical Importance | 35 |
| | | 10.5.1. | Laboratory Values | 35 |
| | | 10.5.2. | ECG | |
| | | 10.5.3. | Vital Signs | 36 |
| | 10.6. | Appendi | x 6: Abbreviations & Trade Marks | 37 |
| | | 10.6.1. | Abbreviations | 37 |
| | | 10.6.2. | Trademarks | 38 |
| | 10.7. | Appendi | x 7: List of Data Displays | 39 |
| | | 10.7.1. | Mock Example Shell Referencing | 39 |
| | | 10.7.2. | Deliverables | |
| | | 10.7.3. | Study Population Tables | 40 |
| | | 10.7.4. | Biomarker Tables | 41 |
| | | 10.7.5. | Biomarker Figures | 44 |
| | | 10.7.6. | ICH Listings | 49 |
| | | 10.7.7. | Non-ICH Listings | |
| | 10.8. | Appendi | x 8: Example Mock Shells for Data Displays | |

#### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the safety and biomarker analyses required for dose escalations and planned biomarker analyses required for interim analyses for Protocol:

| Revision Chronology | Revision Chronology: | |
|---|---|---|
| 2016N309726_00 | 08-May-2017 | Original |
| 2016N309726_01 | 07-AUG-2017 | Change of GM-CSF (LEUKINE) administration from subcutaneous to IV infusion. This is due to liquid LEUKINE no longer being available from the manufacturer Sanofi-Aventis, however lyophilised LEUKINE is available. The guidelines for reconstitution of lyophilised LEUKINE prevent us from administering by subcutaneous as the volume would be too high. In order to remain consistent with clinical practice in dosing GM-CSF therapeutically the dose will be calculated using body surface area. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 08-May-2017) and protocol amendment 1 (Dated: 07-Aug-2017) are outlined in Table 1 for this version of the RAP.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Considerations | Statistical Analysis Plan | Rationale for Changes |
| Sample size re-estimation will be conducted following Part I of the study. | Sample size re-estimation<br>will not be conducted | The methodology used for the original sample size calculation is no longer applicable, therefore the sample size re-estimation will not be conducted. Instead a set of criteria outlined in Section 3.2 will be used to decide if additional participants will be enrolled in Part II of the study. |
| Randomized Population (All participants who are randomized to receive and are given the treatment (LPS or GM-CSF challenge)) is defined as one of the analysis population. | Randomized Population will not be used for Analysis | The randomized and safety populations have the same definitions. Hence only safety population would be used. |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To compare and define the time course of soluble and cellular inflammatory biomarkers (and urinary prostaglandins for LPS only) following systemic challenge with LPS or GM-CSF in healthy participants Secondary Objectives To compare soluble and cellular | <ul> <li>For LPS only: time course and magnitude of upregulation of circulating TNF-α and IL-6 as well as urinary tetranor PGDM</li> <li>For GM-CSF only: time course and magnitude of upregulation of circulating total leukocyte numbers.</li> <li>Secondary Endpoints</li> <li>Soluble inflammatory biomarkers in skin blisters (may</li> </ul> |
| inflammatory biomarkers in cantharidin-induced skin blisters at baseline versus systemic challenge with LPS or GM-CSF in healthy participants | <ul> <li>include but not limited to IL-1b, IL-2, IL-6, IL-8, IFNg, TNF-α, MCP-1, GM-CSF, CRP).</li> <li>Blister volumes and differential cell counts (cellular activation markers may include, but not limited to expression of CD16, CD86, CD80, CD163, CD206, CD83, CD40, CD209, HLA-DR in blister leukocytes)</li> </ul> |
| To define the time course of<br>circulating soluble and cellular<br>inflammatory biomarker upregulation<br>following systemic challenge with LPS<br>or GM-CSF in healthy participants | Time course of regulation of circulating leukocyte numbers and cellular activation markers (may include, but not limited to expression of CD16, CD86, CD80, CD163, CD206, CD83, CD40, CD209, HLA-DR in circulating leukocytes) |
| Exploratory Objectives | Exploratory Endpoints |
| To compare suitability of blisters<br>sampled at 24 and 48 hours <sup>[2]</sup> after<br>induction for maximising observed<br>effects of systemic challenge | <ul> <li>Primary and Secondary endpoints measured in 24 versus<br/>48 hour blisters</li> </ul> |
| To assess the safety and tolerability<br>profile of the challenge agents and to<br>ensure it is not materially different<br>from previous experience. | Adverse events, clinical laboratory measures, vital signs, pain scale assessments |
| Determining whether carboxyesterase-1 (CES-1) expression is present in monocytes following systemic GM-CSF challenge | Number of monocytes which are CES-1+ in blood |
| To compare prostaglandins in urine,<br>blister fluid and plasma at baseline<br>versus systemic challenge with LPS<br>or GM-CSF | Quantification of prostaglandins including (but not limited to [3]) tetranor -PGDM, tetranor-PGEM, PGD2 and PGE2 |
| To assess changes in whole blood<br>transcriptome induced by systemic<br>LPS or GM-CSF | Analysis of differential gene expression in whole blood taken pre-challenge and at selected times post- challenge |
| For LPS challenge only: to assess<br>whether the dose of in -vivo LPS<br>challenge is sufficient to induce innate<br>immune tolerance | <ul> <li>Quantification of inflammatory markers including (but not<br/>limited to) TNF-α and IL-6 in blood drawn pre- and 6 hour<br/>post-systemic LPS challenge following ex vivo incubation<br/>in 'LPS-TruCulture' tubes and LPS-null TruCulture'</li> </ul> |


| Objectives | Endpoints |
|---|---|
| | tubes <sup>[3]</sup> |
| To assess the effects of systemic LPS and GM-CSF challenges on blister healing times | Blister healing times (self-reported in participant diary card) |
| <ul> <li>[1] As an exploratory endpoint, samples will be measured in the Somalogics assay.</li> <li>[2] Blister samples will also be used in the Somalogics assay.</li> <li>[3] Protein panels: IL-6, TNF-α (tolerized proteins), GRO-a (CXCL1) (unchanged) &amp; IL-8 &amp; IL-10 (hyper-responsive)</li> </ul> | |

# 2.3. Study Design



| Overview of St | Overview of Study Design and Key Features |
|---|---|
| Features | <ul> <li>For Part I, a dose exploration design is used to find a dose that provides a robust inflammatory response for both LPS and GM-CSF.</li> <li>For Part II, an additional cohort of up to 8 participants may be enrolled if an interim analysis indicates that this would provide further precision on estimates of primary endpoints. The same 2-session design, as described above, would be used and participants will be dosed with LPS and GM-CSF at the same dose as the 8 evaluable participants from Part I.</li> </ul> |
| Time & Events | Refer to Appendix 1: Schedule of Activities |
| Treatment<br>Assignment | <ul> <li>Participants will be randomised to receive either a LPS or GM-CSF in vivo challenge.</li> <li>The total study duration for each participant is approximately 13 weeks from screening to the final follow-up.</li> </ul> |
| Interim<br>Analysis | <ul> <li>There will be ongoing data reviews conducted by the study team of any available data through the study progression.</li> <li>For Part I, data reviews will be performed by the study team to support whether to dose escalate to the next cohort for each challenge agent.</li> <li>At the end of Part 1, an interim analysis will be conducted to decide whether to enrol additional participants in Part II of the study, for the optimum dose selected in Part I.</li> </ul> |

# 2.4. Statistical Hypotheses / Statistical Analyses

This is an exploratory enabling study which is primarily designed to estimate the effect of systemic exposure to LPS or GM-CSF challenge on soluble and cellular inflammatory biomarkers in blood, urine and cantharidin-induced skin blisters. There are no formal hypotheses to be tested.

# 3. PLANNED ANALYSES

Safety and biomarker data were reviewed on an ongoing basis throughout the progression of the study for dose escalation.

# 3.1. Dose Escalation

| Dose<br>Escalation | Details |
|---|---|
| Study<br>Review<br>Committee<br>(SRC) | <ul> <li>Core GSK members included:</li> <li>Study Physician Lead or their delegate; SERM; Statistician; Operations Study Lead; Epigenetics DPU, MM DPU, Scientific Operations Director, Clinical Development Manager.</li> </ul> |
| Timing | <ul> <li>For each challenge agent, when 2 participants were dosed (n=2 with LPS, n=2 with GM-CSF), a dose escalation meeting was held to make an assessment of tolerability and inflammatory response from Cohort 1.</li> <li>The dose escalation meeting was held prior to Group A in Cohort 2 being dosed with the challenge agents in Session 2.</li> <li>The dose escalation procedure was continued until a well-tolerated dose for LPS and GM-CSF showing a robust inflammatory response was identified.</li> </ul> |
| Safety Data<br>Required | <ul> <li>Ongoing safety data was reviewed, these included: <ul> <li>Participant clinical parameters (including pulse, blood pressure, respiratory rate, temperature &amp; ECG)</li> <li>Adverse events experienced by participants</li> <li>A physician's clinical assessment of participant's tolerability of the prior dose of GM-CSF or LPS with presence (or absence) of symptomatic tachycardia, symptomatic hypo- or hypertension, pyrexia &gt; 38.5c, vomiting, meningeal symptoms, rigors and any other symptoms of concern</li> <li>Review of safety blood tests including FBC (and differential), U&amp;E, CRP, LFT, glucose</li> <li>Other clinical features which in the judgement of the attending physician was pertinent to dose escalation decisions</li> </ul> </li> <li>Safety data was provided from PIMS (i.e. summaries and/or listings).</li> </ul> |
| Biomarker<br>Data<br>Required | <ul> <li>Primary endpoints (across all time points) were reviewed:</li> <li>LPS: Circulating plasma levels of TNF-α and IL-6 as well as urinary tetranor PGDM.</li> <li>GM-CSF: Circulating total leukocyte numbers.</li> <li>Other available data were also reviewed to support dose escalation, but were not formally included in any dose escalation decision criteria:</li> <li>MSD &amp; ELISA readouts from plasma, ex-vivo stimulations and blister fluid samples, Flow Cytometry readouts from blood and blister fluid / blister cell counts.</li> <li>Raw data for biomarkers specified were reviewed (i.e. raw data from GSK CUC</li> </ul> |

| Dose<br>Escalation | Details |
|---|---|
| | included: MSD/ELISA/Flow & TDL (cell counts) and raw data from GSK BIB group for urinary tetranor PGDM.) |
| Statistical<br>Analyses | There were no planned formal statistical analyses of the data. Graphs were created in Excel based on the raw data obtained (nonstandard) |
| Dose<br>Escalation<br>Criteria | Below is the Dose Escalation Criteria decided by the study team If only one participant hits stopping criteria then there will be a presumption of stopping escalation, unless in the judgement of the team further escalation would provide additional scientific value to the study without materially impacting on participant wellbeing. |
| | LPS: STOP dose escalation, IF: |
| | <ul> <li>Peak plasma/serum level of TNF-α ≥ 100 pg/mL (minimum increase of 75 pg/ml from baseline) AND</li> </ul> |
| | <ul> <li>Peak plasma/serum level of IL-6 ≥ 200 pg/mL (minimum increase of 100 pg/ml from baseline) AND</li> </ul> |
| | Urinary tetranor PGDM 3x over baseline in urine OR |
| | <ul> <li>Presence of adverse clinical signs (fever, HR + others) which, in the opinion of<br/>the investigator, pose an unacceptable risk to participants were dose<br/>escalation to proceed. Examples may include, but are not limited to: <ul> <li>Rigors</li> </ul> </li> </ul> |
| | <ul> <li>Meningeal symptoms of moderate severity</li> <li>Vomiting</li> </ul> |
| | <ul> <li>Clinically significant hypotension, hypertension, tachycardia or bradycardia</li> <li>GM-CSF: STOP dose escalation IF:</li> </ul> |
| | <ul> <li>Max change of circulating total leukocyte counts increase by 5 giga/L OR</li> <li>Presence of adverse clinical signs (fever, HR + others) which, in the opinion of the investigator, pose an unacceptable risk to participants were dose escalation to proceed. Examples may include, but are not limited to: <ul> <li>Rigors</li> </ul> </li> </ul> |
| | <ul> <li>Meningeal symptoms of moderate severity</li> </ul> |
| | <ul> <li>Vomiting</li> </ul> |
| | <ul> <li>Clinically significant hypotension, hypertension, tachycardia or<br/>bradycardia</li> </ul> |
| | Elevation of platelet count above 500 x 10 <sup>9</sup> /L |
| Dose<br>Escalation | Following each dose escalation meeting, the decision to STOP or dose escalate for each challenge agent was documented, |
| Decision | <ul> <li>An optimum dose of 0.75 ng/kg for LPS and 60 ug/m2 for GM-CSF was<br/>identified.</li> </ul> |

# 3.2. Interim Analyses

| Interim<br>Analysis | Details |
|---|---|
| Study<br>Review<br>Committee | <ul> <li>Core GSK members include:</li> <li>Study Physician Lead or their delegate; SERM; Statistician; Operations Study Lead; Epigenetics DPU, MM DPU, Scientific Operations Director, Clinical Development Manager.</li> </ul> |
| Timing | At the end of Part I, an interim analysis will be conducted to decide whether to enrol additional participants in Part II of the study, for the optimum dose of 0.75 ng/kg for LPS and 60 ug / m2 for GM-CSF selected in Part I. |
| Biomarker<br>Data<br>Required | <ul> <li>Data for Biomarkers listed in Section 10.3.3 will be presented in tabular and<br/>graphical format and summarized descriptively according to GSK's IDSL<br/>standards.</li> </ul> |
| Statistical<br>Analyses | There are no planned formal statistical analyses of the data. Descriptive summaries and/or graphical presentations will be presented, including data listings. |
| Criteria for<br>Part II | If at least one participant meets the criteria below for the optimal dose of 0.75ng/kg for LPS challenge or 60 ug/m2 for GM-CSF challenge, then Part II of the study will be initiated. Participants will be enrolled to Part II – LPS Challenge at the dose level |
| | 0.75 ng/kg if for at least one participant: |
| | <ul> <li>Maximum increase from baseline at any timepoint in plasma level of TNF-α</li> <li>&lt; 50 pg/mL AND</li> </ul> |
| | <ul> <li>Maximum increase from baseline at any timepoint in plasma level of IL-6 &lt; 50 pg/mL AND</li> </ul> |
| | Maximum increase from baseline at any timepoint in urinary tetranor PGDM level < 1.3x |
| | Participants will be enrolled to Part II – GM-CSF Challenge at the dose level 60 ug/m2 if for at least one participant: |
| | <ul> <li>Maximum increase from baseline at any timepoint in total leukocyte counts &lt;</li> <li>5 giga/L</li> </ul> |
| | Note: Available data from all biomarkers will be considered before making the decision to move to Part II – GM-CSF Challenge. |
| Part II<br>Decision | The decision to STOP after Part I or CONTINUE to Part II for each challenge agent will be documented, including any supporting data. |
| Biomarkers<br>for Part II | If a decision is made to continue to Part II of the study, then biomarkers meeting the criteria below will not be assessed in Part II. |
| | RNASeq and Somalogics data will not be collected for participants in Part II. |
| | If any biomarker is not detectable (< LLQ) at all timepoints for all participants |

| Interim<br>Analysis | Details |
|---|---|
| | of Part I at the optimal dose, the biomarker will not be assessed in Part II. |
| | <ul> <li>If all analytes collected from a single sample type are not detectable (<llq) all="" at="" be="" collected="" dose,="" for="" i="" ii.<="" in="" li="" not="" optimal="" part="" participants="" sample="" the="" then="" this="" timepoints="" will=""> </llq)></li></ul> |
| | <ul> <li>Additionally, the available data for all biomarkers of Part I will be reviewed to<br/>help decide if the biomarkers need to be assessed in Part II.</li> </ul> |

If the decision is made to Stop after Part I, then the RAP for the Final Reporting will follow and additional displays will be generated as part of the Final Reporting.

# 3.3. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for releasing the randomization codes have been met (where required).
- 4. Randomization codes have been distributed according to RandAll NG procedures.

## 4. ANALYSIS POPULATIONS

| Population | Definition /Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | <ul> <li>Selected Study<br/>Population</li> </ul> |
| Enrolled | <ul> <li>All participants who passed screening and entered the study. Included are: Run-in Failures; Randomized Participants; in non-randomized study and participants who were assigned a treatment in a non-randomised study.</li> <li>Note screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study.</li> </ul> | Selected Study<br>Population |
| Safety | <ul> <li>All participants who are randomized to receive the treatment (LPS or GM-CSF challenge) and received at least one dose of challenge agent.</li> <li>This population will be based on the challenge agent participants actually received.</li> <li>Note: Participants who were not randomized but received at least one dose of challenge agent should be listed.</li> </ul> | <ul><li>Biomarker</li><li>Safety</li></ul> |

<sup>[1]</sup> Refer to Appendix 7: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed as part of the Final Reporting.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan [06Feb2018 V1.1] or higher.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF. For the Interim Analysis, no displays related to protocol deviations and inclusion/exclusion criteria deviations will be generated.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description | Order in TLF |
| Α | LPS Dose 1 | LPS 0.5 ng/kg | 1 |
| В | LPS Dose 2 | LPS 1.0 ng/kg | 3 |
| С | LPS Dose 3 | LPS 0.75 ng/kg | 2 |
| D | LPS Dose 4 | LPS 0.75 ng/kg | 2 |
| G | GM-CSF Dose 1 | GM-CSF 60 ug/m2 | 4 |
| Н | GM-CSF Dose 2 | GM-CSF 60 ug/m2 | 4 |

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose of challenge and used as baseline.

| Parameter | Study As | ssessments ( | Baseline Used in Data | | |
|---|---|---|---|---|---|
| | Screening | Session 1<br>Day 1 | Session 1<br>Day 2 | Session 2<br>Day 1 | Display |
| Biomarkers | | | | | |
| LPS: TNF-α, IL6<br>GM-CSF: WBC (Total<br>leukocyte counts) | | X | X | X | Session 2 Day 1 (Pre<br>Blister Induction) |
| Blood | | Х | | | Session 1 Day 1 (Pre<br>Blister Induction) |
| Blister | | | Х | | Session 1 Day 2<br>(24 HR) |
| Urine | | | Χ | | Session 1 Day 2 (Pre Fluid Sampling) |
| In Vivo LPS or GM-CSF | | | | X | Session 2 Day 1 (Pre<br>Blister Induction) |
| Safety | | | | | |
| Vital Signs &<br>Temperature | Х | Х | | | Session 1 Day 1 |
| ECG | Х | | | | Screening |
| Labs | Χ | Х | | | Session 1 Day 1 |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Examination of Covariates, Other Strata and Subgroups

#### 5.3.1. Covariates and Other Strata

There are no planned covariates or other strata that will be used in descriptive summaries and statistical analyses, if conducted.

## **5.3.2.** Examination of Subgroups

There are no planned sub-group analyses.

# 5.4. Multiple Comparisons and Multiplicity

Analyses, if conducted will not be subject to any multiplicity adjustment.

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions for Interim Reporting are outlined in the appendices:

| Section | Component |
|---------|-----------------------------------------------------------|
| 10.2 | Appendix 2: Data Display Standards & Handling Conventions |
| 10.3 | Appendix 3: Derived and Transformed Data |
| 10.4 | Appendix 4: Reporting Standards for Missing Data |
| 10.5 | Appendix 5: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Enrolled" population, unless otherwise specified. Screen failures will be listed based on the "Screened" population.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK IDSL Data Standards. Details of the planned displays are presented in Appendix 7: List of Data Displays.

For the Interim Analysis, only a Summary and Listing of Demographic Characteristics will be presented.

#### 7. EFFICACY ANALYSES

## 7.1. Primary Biomarker Analyses

Unless otherwise stated, analyses will apply to the interim analyses.

#### 7.1.1. Endpoint / Variables

| Challenge | Endpoint |
|---|---|
| LPS | Time course and magnitude of upregulation of circulating TNF- $\alpha$ and IL-6 as well as urinary tetranor PGDM |
| GM-CSF | Time course and magnitude of upregulation of circulating total leukocyte numbers. |

## 7.1.2. Summary Measure

| Challenge | Endpoint |
|---|---|
| LPS | Absolute values and change from baseline in TNF-α, IL-6 and PGDM across the |
| | time course |
| | Baseline: |
| | <ul> <li>TNF-α, IL-6: Session 2: Day 1 (Pre Blister Induction)</li> </ul> |
| | PGDM: Session 1 Day 2 (Pre Fluid Sampling) |
| GM-CSF | Absolute values and change from baseline in total leukocyte across the time course |
| | Baseline = Session 2: Day 1 (Pre Blister Induction) |

# 7.1.3. Population of Interest

The primary biomarker analyses will be based on the "Safety" population, unless otherwise specified.

# 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

No Strategy for Intercurrent (Post-Randomization) Events has been planned for this study.

## 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 7: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.2. Secondary Biomarker Analyses

Unless otherwise stated, analyses will apply to the interim analyses.

#### 7.2.1. Endpoint / Variables

There are several different types of biomarker samples collected during the study:

- Biomarkers from skin blister fluid (i.e. mediators and flow cytometry)
- Biomarkers from blood sample (i.e. mediators, flow cytometry, ex vivo stimulation (LPS only) and transcriptome)
- Biomarkers from urine (Primary endpoints)

The secondary endpoints of interest with respect to the biomarkers mentioned above:

#### **Endpoint**

Soluble and cellular inflammatory biomarkers in cantharidin-induced skin blisters at baseline versus systemic challenge with LPS or GM-CSF in healthy participants

Time course of circulating soluble and cellular inflammatory biomarker upregulation

#### 7.2.2. Summary Measure

Absolute values and change from baseline of soluble and cellular inflammatory biomarkers across the time course.

Note: In the Interim Analysis, for the biomarkers from skin blister fluid, values will be averaged across arms (left and right) for each participant. These averaged values will be used in tables and figures.

If one of the values is not collected or is missing, then the single value present in the data will be used in tables and figures. Appropriate footnotes will be provided to reflect data are not an average value.

#### 7.2.3. Population of Interest

The secondary biomarker analyses will be based on the "Safety" population, unless otherwise specified.

#### 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

No Strategy for Intercurrent (Post-Randomization) Events has been planned for this study.

## 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 7: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.3. Exploratory Biomarker Analyses

#### SomaLogic

- The full panel of analytes contains 1305 proteins, and these will be measured from 88 plasma samples and 32 blister samples.
- Data will be delivered as relative fluorescense units, in two batches (one for each sample type).
- Data will be viewed as individual proteins and individual donors. This provides
  indication of how proteins change within an individual by reviewing the data.
  However, if effects across participants (i.e. N=4 for LPS or N=4 for GM-CSF) needs
  to be assessed, data will be normalised prior to analyses.
- Data will only be analysed at the end of the study as part of the Final Reporting.
   Further considerations for analysis will be detailed in the RAP as part of the Final Reporting.

#### **RNA Seq Data**

RNAseq data will provided by Expression Analysis at Q Squared Solutions in a
FASTQ file format. Data in this format will be directly analysed by GSK
Computational biology groups. Analysis summary files containing summaries of
information such of alignment statistics, mapping quality, base distributions, most
frequent gene detected and total number of genes, by sample, will be generated.
RNAseq will be analysed outside this reporting effort.

# 8. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified. There are no Safety Analyses planned for the Interim.

# 9. REFERENCES

GlaxoSmithKline Document Number 2016N309726\_01 Study ID 207654: An open label parallel group study to investigate the optimum methodology for the use of LPS or GM-CSF as challenge agents on healthy participants by assessing inflammatory biomarkers in cantharidin-induced skin blisters, peripheral blood, and urine.

Effective Date: 07-AUG-2017

# 10. APPENDICES

# 10.1. Appendix 1: Schedule of Activities

# 10.1.1. Protocol Defined Schedule of Events

| PROCEDURE Day: | Screening | S | ESSION | 11 | Interim<br>inspection | | | | 7000 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Within 30<br>days of<br>Day 1 | Day<br>1 | Day<br>2 | Day<br>3 | Minimum<br>2 wks<br>(max 4<br>weeks)<br>after end<br>of session | Day<br>-1 | Day<br>1 | Day<br>2 | Day<br>3 | Minimum<br>2 wks (max. 4<br>weeks) after<br>end of<br>session 2 | Approx.<br>5wks after<br>end of<br>session 2 | | |
| Attend Unit | Χ | X | Χ | Χ | X | Х3 | X3 | Χ | Х | X | X | 1. | Brief physical exam only |
| Informed Consent | X | | | | | | | | | | | 2. | Within an hour before |
| Inclusion/Exclusion checklist | X | | | | | Х | | | | | | | cantharidin application |
| Medical /medication history | X | | | | | | | | | | | 3. | Overnight stay in the unit |
| Demographics | X | | | | | | | | | | | 4. | Additional clinical lab |
| Body weight | X | | | | | X | | | | | | ì | assessments may be |
| Drug/alcohol test | X | X | | | | X | | | | | | | performed, if necessary |
| Physical Exam | X | X1 | | | | Х | X1 | | | X1 | 31150 | 5.<br>6 | Before blister fluid sampling<br>After the last blister fluid |
| Vital Signs and temperature | Х | X <sup>2</sup> | | | | Х | X8 | X | | X | X | 0. | sampling at each session |
| ECG | X | | | | | Х | X | | | | | 7. | Multiple blood draws at the |
| Telemetry | | | | | | 88 · | X | | | | | | following time points: Pre |
| Visual forearm check<br>(including blister healing and<br>cosmetic assessment) | Х | X2 | | | X | Х | X <sup>2</sup> | | | X | X | | challenge, ,<br>5 mins (i.e. Pre-blister<br>induction), 10 min, 25 min, 40 |
| Cantharidin application<br>(Session 2 only: 20 minutes<br>post end of LPS or GM-CSF<br>challenge) | | X | | | | | X | | | | | | min, 1hr:10mins, 1hr:40mins,<br>2hr:40mins, 5hr:40mins with<br>respect to start of blister<br>induction |
| | | | | | | | | | | 8. | Every half hour for the first 4 | | |
| SAE | «- | | | | | | | | | | » | | hours after challenge, hourly |
| Clinical Chemistry,<br>Haematology, and Urinalysis | Х | X | X | X | | Х | Х | X | Х | | | | until 8 hours and then 8 hourly<br>until discharge. Frequency can<br>be increased if symptomatic |
| Mediators blood sample | | X <sup>2</sup> | X5 | χ5 | | Ü | X7 | X5 | X5 | | | 9. | For flow cytometry and |
| Flow cytometry blood sample | | X2 | χ5 | χ5 | 10 | | X9 | X5 | χ5 | | | | transcriptomic blood samples: |
| For LPS only: Ex vivo | | | | | | | X10 | | | | | 1 | Multiple blood draws at the |

| PROCEDURE | Screening | SI | ESSION | 11 | Interim<br>inspectio<br>n | | SESS | SION 2 | | 1st<br>follow-up | 2nd<br>follow-up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day: | Within 30<br>days of<br>Day 1 | Day<br>1 | Day<br>2 | Day<br>3 | Minimum<br>2 wks<br>(max 4<br>weeks)<br>after end<br>of session | Day<br>-1 | Day<br>1 | Day<br>2 | Day<br>3 | Minimum<br>2 wks (max. 4<br>weeks) after<br>end of<br>session 2 | Approx.<br>5wks after<br>end of<br>session 2 | | |
| stimulation blood sample | | | | | | | | | | | | | following time points: Pre |
| Transcriptomic blood sample | | | | | | | Х9 | | | | | | challenge, 40 mins, 2hr:40mins |
| Urine sampling for PD | | | X11 | | | | X11 | | | | | | and 5hr:40mins (and 9hr |
| For LPS only: Intravenous hydration with normal Saline | | | | | | | X12 | | | | | | 40mins for GM-CSF for flow<br>cytometry only) with respect to<br>start of blister induction |
| at a rate of 250 mL / hr<br>In vivo I PS or GM-CSF | | | | | | | X2 | - | | | | 10 | Ex vivo stimulation blood |
| challenge | | | | | | | λ2 | , | | 5 | | 10. | sample: 2 samples (one null<br>and one LPS tube) to be taken |
| Blister sample for biomarkers | | | X | Χ | | | | Х | Χ | | | | |
| Pain rating <sup>6</sup> Participant diary card given to participant to record blister healing | | Х | | X | | | X | | X | | | 11. F | pre-dose and 2 samples (one null and one LPS tube) to be taken at 5hrs:40mins post blister induction Pre-challenge urine sample will be collected in session 1. For the post-challenge samples in session 2, participants will be encouraged to pass urine immediately before LPS dosing and each urine void will be collected after LPS until 12 hours post-LPS From 4 hours prior to LPS until 8 hours after LPS |

# 10.2. Appendix 2: Data Display Standards & Handling Conventions

## 10.2.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | HARP Server : UK1SALX00175 |
| HARP Compound | HARP Compound : NOCOMPOUND\MID207654\Internal_01 |
| Analysis Datasets | |
| Analysis datasets will be created per GSK IDSL dataset standards. | |
| Generation of RTF Files | |
| RTF files will be generated for interim reporting effort. | |

## 10.2.2. Reporting Standards

#### General

The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless
otherwise stated

(IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- All displays will use the term "Subject", the term "Subject" is used to refer to a participant in the protocol.
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
  - For all Biomarkers, the following DP's places will be applied:
  - Summary Statistics: Maximum of 4 DP's for Mean and Median, 5 DP's for SD, 3 DP's for Min and Max.
  - Listings: Provide DP's in BEST. format.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL)


| Statistical Prin | Statistical Principle 5.05.1). |
|---|---|
| <ul> <li>Unscheduled</li> </ul> | <ul> <li>Unscheduled or unplanned readings will be presented within the subject's listings.</li> </ul> |
| <b>Unscheduled Visits</b> | Unscheduled Visits |
| Unscheduled visits | Unscheduled visits will not be included in summary tables and/or figures. |
| All unscheduled vi | All unscheduled visits will be included in listings. |
| Descriptive Summary | Descriptive Summary Statistics |
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data N, n, frequency, % | |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

#### 10.3. Appendix 3: Derived and Transformed Data

#### 10.3.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.
- For the biomarkers from skin blister fluid, values will be averaged across arms (left and right) for each
  participant. These averaged values will be used in tables and figures. If one of the values is not
  collected or is missing, then the single value present in the data will be used in tables and figures.
  Appropriate footnotes will be provided to reflect data are not an average value.

#### Study Day

- Calculated as the number of days from Challenge Administration Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Challenge Administration Date → Study Day = Ref Date Challenge Administration
    Date</li>
  - Ref Data ≥ Challenge Administration Date → Study Day = Ref Date (Challenge Administration Date) + 1

## 10.3.2. Study Population

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
- Any participant with a missing day will have this imputed as day '15'.
- Any participant with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- If only birth year is collected, then the birth date and month will be imputed as '30th June' for calculating age.
- The reference day for age calculation will be screening visit.

#### 10.3.3. Biomarker

The table below provides the list of Biomarkers needed for Interim.

Biomarker Code (BICATCD), Biomarker Test Code (BITESTCD), Biomarker Testing Method Code (BIMETHCD) and Units of Measurement (BIORRESU) can be referred below.

| Name<br>(Analyte) | Biomarker Detailed Name | BICATCD | BITESTCD/<br>BIMETHCD/<br>BIORRESU |
|---|---|---|---|
| Soluble<br>Inflammatory<br>Mediators | Tumour necrosis factor alpha (TNF-α) | TNFA | CONC/<br>MSD/<br>PG/ML |
| (Blood)<br>Primary | Interleukin 6 | IL6 | CONC/<br>MSD/<br>PG/ML |
| Soluble<br>Inflammatory<br>Mediators | C-reactive protein (LAB dataset) Monocyte chemotactic | LBTESTCD:<br>CRP_PLC<br>MCP1 | LBORUNIT:<br>MG/L<br>CONC/ |
| (Blood)<br>Secondary | protein-1 | | MSD/<br>PG/ML |
| | Monocyte chemotactic protein-4 | MCP4 | CONC/<br>MSD/<br>PG/ML |
| | Eotaxin | EOTAXIN | CONC/<br>MSD/<br>PG/ML |
| | Inducible protein 10 | IP10 | CONC/<br>MSD/<br>PG/ML |
| | MDC | MDC | CONC/<br>MSD/<br>PG/ML |
| | Chemokine (C-C motif) ligand 26 gene | CCL26 | CONC/<br>MSD/<br>PG/ML |
| | Thymus and activation-<br>regulated chemokine | TARC | CONC/<br>MSD/<br>PG/ML |
| | Macrophage inflammatory protein 1 alpha | MIP1A | CONC/<br>MSD/<br>PG/ML |
| | Macrophage inflammatory protein 1 beta | MIP1B | CONC/<br>MSD/<br>PG/ML |
| | Interferon-gamma | IFNG | CONC/<br>MSD/<br>PG/ML |
| | Interleukin 10 | IL10 | CONC/<br>MSD/<br>PG/ML |
| | Interleukin 12 p70 | IL12P70 | CONC/<br>MSD/<br>PG/ML |

| Name | Biomarker Detailed Name | BICATCD | BITESTCD/ |
|---|---|---|---|
| (Analyte) | | | BIMETHCD/ |
| | | | BIORRESU |
| | Interleukin 1 beta | IL1B | CONC/ |
| | | | MSD/ |
| | | | PG/ML |
| | Interleukin 8 | IL8 | CONC/ |
| | | | MSD/ |
| | | | PG/ML |
| | Activin-A | ACTIVA | CONC/ |
| | | | ELISA/ |
| | | | PG/ML |
| | Matrix metalloproteinase-1 | MMP1 | CONC/ |
| | (interstitial collagenase) | | MSD/ |
| | | | PG/ML |
| | Matrix metalloproteinase 3 | MMP3 | CONC/ |
| | | | MSD/ |
| | | | PG/ML |
| | Matrix metalloproteinase 9 | MMP9 | CONC/ |
| | | | MSD/ |
| | | | PG/ML |
| | Granulocyte macrophage | GMCSF | CONC/ |
| | colony stimulating factor | | ELISA/ |
| 0.1.1. | | 11.40 | PG/ML |
| Soluble | Interleukin 10 | IL10 | CONC/ |
| Inflammatory | | | MSD/ |
| Mediators | Interior C | IL6 | PG/ML |
| (Blood -<br>TruCulture) | Interleukin 6 | ILO | CONC/<br>MSD/ |
| Truculture) | | | PG/ML |
| | Interleukin 8 | IL8 | CONC/ |
| | Interieukin o | ILO | MSD/ |
| | | | PG/ML |
| | Tumour necrosis factor alpha | TNFA | CONC/ |
| | (TNF-α) | TINIA | MSD/ |
| | (1111 3) | | PG/ML |
| | Chemokine (C-X-C motif) | CXCL1 | CONC/ |
| | ligand 1 (melanoma growth | 07.02. | ELISA/ |
| | stimulating activity, alpha) | | PG/ML |
| Soluble | Monocyte chemotactic | MCP1 | CONC/ |
| Inflammatory | protein-1 | | MSD/ |
| Mediators | | | PG/ML |
| (Blister) | Interleukin 10 | IP10 | CONC/ |
| | | | MSD/ |
| | | | PG/ML |
| | Thymus and activation- | TARC | CONC/ |
| | regulated chemokine | | MSD/ |
| | | | PG/ML |

| Name | Biomarker Detailed Name | BICATCD | BITESTCD/ |
|---|---|---|---|
| (Analyte) | | | BIMETHCD/<br>BIORRESU |
| | Interleukin 12 p70 | IL12P70 | CONC/<br>MSD/ |
| | Activin-A | ACTIVA | PG/ML CONC/ ELISA/ |
| | Matrix metalloproteinase-1 (interstitial collagenase) | MMP1 | PG/ML CONC/ MSD/ PG/ML |
| | Matrix metalloproteinase 3 | MMP3 | CONC/<br>MSD/<br>PG/ML |
| | Matrix metalloproteinase 9 | MMP9 | CONC/<br>MSD/<br>PG/ML |
| Soluble<br>Inflammatory<br>Mediators | Tetranor-Prostaglandin E<br>Metabolite | TETPGDM | CONC/<br>LCMS/<br>PG/ML |
| (Urine)<br>Primary | Tetranor-Prostaglandin D<br>Metabolite | TETPGEM | CONC/<br>LCMS/<br>PG/ML |
| Cell Numbers<br>(Blood)<br>Primary | White blood cells | WBC | TNCELL/ FLWCY/<br>CELLS/ML |
| Blister Volume<br>(Blister) | Blister Fluid | BLISTFL | VOL/<br>WTDENC/<br>UL |
| Flow<br>Cytometry | CD16+ | CD16 | C6/<br>FLWCY/<br>MNFI |
| Cell Activation<br>Markers on<br>Monocytes | CD86+ | CD86 | C6/<br>FLWCY/<br>MNFI |
| (Blister and<br>Blood) | CD80 molecule | CD80 | C6/<br>FLWCY/<br>MNFI |
| | CD163+ | CD163 | C6/<br>FLWCY/<br>MNFI |
| | CD206+ | CD206 | C6/<br>FLWCY/<br>MNFI |
| | CD83 molecule | CD83 | C6/<br>FLWCY/<br>MNFI |

| Name<br>(Analyte) | Biomarker Detailed Name | BICATCD | BITESTCD/<br>BIMETHCD/<br>BIORRESU |
|---|---|---|---|
| | CD40 | CD40 | C6/<br>FLWCY/<br>MNFI |
| | CD209+ | CD209 | C6/<br>FLWCY/<br>MNFI |
| | HLA-DR | HLADR | C6/<br>FLWCY/<br>MNFI |
| | CD40+/CD80+ | CDX690 | %MONO/<br>FLWCY/<br>% |
| Flow<br>Cytometry | CD16+ | CD16 | R1/<br>FLWCY/<br>MNFI |
| Cell Activation Markers on Dendritic Cells | CD86+ | CD86 | R1/<br>FLWCY/<br>MNFI |
| (Blister and Blood) | CD80 molecule | CD80 | R1/<br>FLWCY/<br>MNFI |
| | CD163+ | CD163 | R1/<br>FLWCY/<br>MNFI |
| | CD206+ | CD206 | R1/<br>FLWCY/<br>MNFI |
| | CD83 molecule | CD83 | R1/<br>FLWCY/<br>MNFI |
| | CD40 | CD40 | R1/<br>FLWCY/<br>MNFI |
| | CD209+ | CD209 | R1/<br>FLWCY/<br>MNFI |
| | HLA-DR | HLADR | R1/<br>FLWCY/<br>MNFI |
| | CD40+/CD80+ | CDX690 | %TDC/<br>FLWCY/<br>% |
| Flow<br>Cytometry | Neutrophils | NEUT | TNCELL/<br>FLWCY/<br>CELLS/ML |

| Name<br>(Analyte) | Biomarker Detailed Name | BICATCD | BITESTCD/<br>BIMETHCD/<br>BIORRESU |
|---|---|---|---|
| Cell Counts<br>(Blood) | Lymphocytes | LYMPH | TNCELL/<br>FLWCY/ |
| | Monocytes | MONO | CELLS/ML TNCELL/ FLWCY/ CELLS/ML |
| | B Cells | BCELL | TNCELL/ FLWCY/ CELLS/ML |
| | CD45+ CD3- CD56+<br>(NK Cells) | CDX223 | TNCELL/<br>FLWCY/<br>CELLS/ML |
| | CD45+ CD3+ CD56+<br>(NKT Cells) | CDX224 | TNCELL/<br>FLWCY/<br>CELLS/ML |
| | Total T Cells | TTCELL | TNCELL/<br>FLWCY/<br>CELLS/ML |
| | CD4+ | CD4 | TNCELL/<br>FLWCY/<br>CELLS/ML |
| | CD8+ | CD8 | TNCELL/<br>FLWCY/<br>CELLS/ML |
| | CD14+CD16+ Monocytes | CDX469 | TNCELL/<br>FLWCY/<br>CELLS/ML |
| | CD14+CD16- Monocytes | CDX471 | TNCELL/<br>FLWCY/<br>CELLS/ML |
| | CD14-CD16+ Monocytes | CDX611 | TNCELL/<br>FLWCY/<br>CELLS/ML |
| | CD34+ | CD34 | TNCELL/<br>FLWCY/<br>CELLS/ML |
| Flow Cytometry Cell Counts (Blister) | Neutrophils | NEUT | TNCELL/ FLWCY/ CELLS/ML or 10^3 CELLS/BLISTER |
| Note: These biomarkers are measured in 2 units – | Lymphocytes | LYMPH | TNCELL/ FLWCY/ CELLS/ML or 10^3 CELLS/BLISTER |

| Name<br>(Analyte) | Biomarker Detailed Name | BICATCD | BITESTCD/<br>BIMETHCD/<br>BIORRESU |
|---|---|---|---|
| Cells/ml and<br>10^3<br>Cells/Blister | Monocytes | MONO | TNCELL/ FLWCY/ CELLS/ML or 10^3 CELLS/BLISTER |
| | B Cells | BCELL | TNCELL/ FLWCY/ CELLS/ML or 10^3 CELLS/BLISTER |
| | CD45+ CD3- CD56+<br>(NK Cells) | CDX223 | TNCELL/ FLWCY/ CELLS/ML or 10^3 CELLS/BLISTER |
| | CD45+ CD3+ CD56+<br>(NKT Cells) | CDX224 | TNCELL/ FLWCY/ CELLS/ML or 10^3 CELLS/BLISTER |
| | Total T Cells | TTCELL | TNCELL/ FLWCY/ CELLS/ML or 10^3 CELLS/BLISTER |
| | CD4+ | CD4 | TNCELL/ FLWCY/ CELLS/ML or 10^3 CELLS/BLISTER |
| | CD8+ | CD8 | TNCELL/ FLWCY/ CELLS/ML or 10^3 CELLS/BLISTER |
| | CD14+CD16+ Monocytes | CDX469 | TNCELL/ FLWCY/ CELLS/ML or 10^3 CELLS/BLISTER |
| | CD14+CD16- Monocytes | CDX471 | TNCELL/ FLWCY/ CELLS/ML or 10^3 CELLS/BLISTER |


| Name<br>(Analyte) | Biomarker Detailed Name | BICATCD | BITESTCD/<br>BIMETHCD/<br>BIORRESU |
|---|---|---|---|
| | CD14-CD16+ Monocytes | CDX611 | TNCELL/<br>FLWCY/<br>CELLS/ML<br>or 10^3<br>CELLS/BLISTER |

# 10.4. Appendix 4: Reporting Standards for Missing Data

# 10.4.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>As specified in the protocol (Section 5.3), a participant is considered to have completed the study if he/she has completed up to the end of session 2 of the study.</li> <li>If a participant withdraws before the end of session 2 they will be encouraged to return for a follow-up visit as per the schedule of activities.</li> </ul> |
| | • If a participant withdraws before the end of session 2 their data may still be used for analysis, depending on how much data is available. If there is insufficient data for analysis, at the discretion of the study team, this participant will be replaced. |
| | • The end of the study is defined as the date of the last visit of the last participant in the Study (e.g. the second follow up session for the last participant). |
| | All available data from participants who were withdrawn from the study will be listed. |

# 10.4.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing</li> </ul> |
| | data and should be displayed as such. |
| | For Biomarkers, the following will be applied: |
| | <ul> <li>If any value is not quantified and the numeric result is absent as the value is below the<br/>lower limit of quantification, then values will be imputed as half of the LLQ.</li> </ul> |
| | • If any value is below the lower limit of quantification but the numeric result is present, then the numeric values will be used in all displays. |
| | • If any value is above ULQ, such values will be omitted from summaries/figures even if the numeric result is present. These values will only be listed. |
| | <ul> <li>Numeric results of samples which are "Plate failed QC" and "CV&gt;20%" will be used in all<br/>displays.</li> </ul> |
| | <ul> <li>Appropriate footnotes will be provided in Tables and Summaries to indicate that <llq,< li=""> <li>CV&gt;20% and Plate Failed Samples have been used.</li> </llq,<></li></ul> |
| | <ul> <li>The diluted samples of the biomarkers whose value is &gt;ULQ will be re-run and the new<br/>reported values will be used in the final analysis.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.4.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |

# 10.5. Appendix 5: Values of Potential Clinical Importance

# 10.5.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Relative – Low<br>(Multipliers of LLN) | Relative – High<br>(Multipliers of ULN) |
| Hematocrit | Ratio of<br>1 | Male | | 1.02 |
| | | Female | | 1.17 |
| | | $\Delta$ from BL | < -0.075 chang | e from baseline |
| Haemoglobin | g/L | Male | | 1.03 |
| | | Female | | 1.13 |
| | | $\Delta$ from BL | < -25 change | e from baseline |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.81 | |
| Neutrophil Count | x109/ L | | 0.83 | |
| Platelet Count | x10 <sup>9</sup> / L | | 0.67 | |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 0.67 | |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Relative – Low Relative – H | |
| | | | (Multipliers of LLN) | (Multipliers of ULN) |
| Albumin | mmol/L | | 0.86 | |
| Calcium | mmol/L | | 0.91 | 1.06 |
| Creatinine | umol/L | $\Delta$ from BL | | 1.25 |
| Glucose | mmol/L | | 0.71 | 1.41 |
| Magnesium | mmol/L | | 0.63 | 1.03 |
| Phosphorus | mmol/L | | 0.80 | 1.14 |
| Potassium | mmol/L | | 0.86 | 1.10 |
| Sodium | mmol/L | | 0.96 | 1.03 |
| Total CO2 | mmol/L | | 0.86 | 1.14 |

| Liver Function | | | |
|---|---|---|---|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| T. Bilirubin + ALT | μmol/L<br>U/L | High | ≥ 1.5xULN T. Bilirubin ≥ 2x ULN ALT |

# 10.5.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | >450 |
| Absolute PR Interval | msec | <110 | >220 |
| Absolute QRS Interval | msec | <75 | >110 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | >60 |

# 10.5.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-----------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Temperature | degrees C | <35.5 | >37.5 |
| Systolic Blood Pressure | mmHg | <85 | >160 |
| Diastolic Blood Pressure | mmHg | <45 | >100 |
| Heart Rate | bpm | <40 | >110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Temperature | degrees C | Change of 1°C from baseline within four hours | | | |
| Systolic Blood Pressure | mmHg | ≥20 | ≥40 | ≥20 | ≥40 |
| Diastolic Blood Pressure | mmHg | ≥10 | ≥20 | ≥10 | ≥20 |
| Heart Rate | bpm | ≥15 | ≥30 | ≥15 | ≥30 |
# 10.6. Appendix 6: Abbreviations & Trade Marks

## 10.6.1. Abbreviations

| Abbreviation | Description |
|---|---|
| A&R | Analysis and Reporting |
| CI | Confidence Interval |
| CS | Clinical Statistics |
| CP | Clinical Programming |
| CPSSO | Clinical Pharmacology Science and Study Operations |
| CRP | C-reactive protein |
| CSR | Clinical Study Report |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| DPU | Discovery Performance Unit |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| ELISA | Enzyme Linked ImmunoSorbent Assay |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GM-CSF | Granulocyte-Macrophage Colony-Stimulating Factor |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IL | Interleukin |
| LLN | Lower Limit of Normal |
| LLQ | Lower Limit of Quantification |
| LPS | Lipopolysaccharide |
| MCH | Mean Corpuscular Hemoglobin |
| MCP | Monocyte chemoattractant protein |
| MM | Muscle Metabolism |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| PGD2 | Prostaglandin D2 |
| PGE2 | Prostaglandin E2 |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| RNA | Ribonucleic acid |
| SAC | Statistical Analysis Complete |
| TA | Therapeutic Area |
| TNF | Tumour Necrosis Factor |
| TFL | Tables, Figures & Listings |
| ULN | Upper limit of normal |

## 10.6.2. Trademarks

Trademarks of the GlaxoSmithKline Group of Companies

HARP

Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

## 10.7. Appendix 7: List of Data Displays

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 | N/A |
| Biomarker | 2.1 to 2.24 | 2.1 to 2.47 |
| Safety | N/A | N/A |
| Section | List | ings |
| ICH Listings | , | 1 |
| Other Listings | 2 to | 14 |

## 10.7.1. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 8: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Biomarker | BIO_Fn | BIO_T1 | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.7.2. Deliverables

| Delivery [1] | Description |
|--------------|------------------------------------------------|
| IA SAC [1] | Interim Analysis Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

## 10.7.3. Study Population Tables

| Study Pop | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Demograp | Demographic and Baseline Characteristics | | | | |
| 1.1. | Enrolled | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | IA [1] |

## 10.7.4. Biomarker Tables

| Biomarke | r Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Soluble Ir | nflammatory M | ediators | | | |
| 2.1. | Safety | BIO_T1 | Summary of Primary Soluble Inflammatory Mediators in Blood | Page by Treatment and Biomarker | IA [1] |
| 2.2. | Safety | BIO_T1 | Summary of Change from Baseline in Primary Soluble Inflammatory Mediators in Blood | Page by Treatment and Biomarker. | IA [1] |
| 2.3. | Safety | BIO_T1 | Summary of Secondary Soluble Inflammatory Mediators in Blood | Page by Treatment and Biomarker | IA [1] |
| 2.4. | Safety | BIO_T1 | Summary of Change from Baseline in Secondary Soluble Inflammatory Mediators in Blood | Page by Treatment and Biomarker | IA [1] |
| 2.5. | Safety | BIO_T1 | Summary of Soluble Inflammatory Mediators from In-Vitro (un)stimulated Blood Pre and Post In-Vivo LPS Challenge | Page by Treatment and Biomarker | IA [1] |
| 2.6. | Safety | BIO_T1 | Summary of Soluble Inflammatory Mediators in Blister | Page by Treatment and Biomarker | IA [1] |
| 2.7. | Safety | BIO_T1 | Summary of Change from Baseline of Soluble Inflammatory Mediators in Blister | Page by Treatment and Biomarker | IA [1] |
| 2.8. | Safety | BIO_T1 | Summary of Soluble Inflammatory Mediators in Urine following LPS Challenge | Page by Treatment and Biomarker | IA [1] |
| 2.9. | Safety | BIO_T1 | Summary of Change from Baseline of Soluble Inflammatory Mediators in Urine following LPS Challenge | Page by Treatment and Biomarker | IA [1] |
| Total Leul | kocyte Number | 's | | | |
| 2.10. | Safety | BIO_T1 | Summary of Cell Numbers in Blood following GM-CSF Challenge | Page by Treatment and Biomarker | IA [1] |
| 2.11. | Safety | BIO_T1 | Summary of Change from Baseline in Cell Numbers in Blood | Page by Treatment and | IA [1] |

| Biomarker Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | following GM-CSF Challenge | Biomarker | |
| Blister Vo | lume | | | | · |
| 2.12. | Safety | BIO_T1 | Summary of Blister Volume | Page by Treatment | IA [1] |
| Flow Cyto | metry | | | | · |
| 2.13. | Safety | BIO_T1 | Summary of Cell Activation Markers by Flow Cytometry on Monocytes in Blood | Page by Treatment and Biomarker | IA [1] |
| 2.14. | Safety | BIO_T1 | Summary of Change from Baseline in Cell Activation Markers by Flow Cytometry on Monocytes in Blood | Page by Treatment and Biomarker | IA [1] |
| 2.15. | Safety | BIO_T1 | Summary of Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blood | Page by Treatment and Biomarker | IA [1] |
| 2.16. | Safety | BIO_T1 | Summary of Change from Baseline in Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blood | Page by Treatment and Biomarker | IA [1] |
| 2.17. | Safety | BIO_T1 | Summary of Cell Counts by Flow Cytometry in Blood | Page by Treatment and<br>Biomarker | IA [1] |
| 2.18. | Safety | BIO_T1 | Summary of Change from Baseline in Cell Counts by Flow Cytometry in Blood | Page by Treatment and Biomarker | IA [1] |
| 2.19. | Safety | BIO_T1 | Summary of Cell Activation Markers by Flow Cytometry on Monocytes in Blister | Page by Treatment and Biomarker | IA [1] |
| 2.20. | Safety | BIO_T1 | Summary of Change from Baseline in Cell Activation Markers by Flow Cytometry on Monocytes in Blister | Page by Treatment and Biomarker | IA [1] |
| 2.21. | Safety | BIO_T1 | Summary of Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blister | Page by Treatment and<br>Biomarker | IA [1] |
| 2.22. | Safety | BIO_T1 | Summary of Change from Baseline in Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blister | Page by Treatment and<br>Biomarker | IA [1] |
| 2.23. | Safety | BIO_T1 | Summary of Cell Counts by Flow Cytometry in Blister | Page by Treatment and | IA [1] |

| Biomarker Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | | Biomarker | |
| 2.24. | Safety | BIO_T1 | Summary of Change from Baseline in Cell Counts by Flow Cytometry in Blister | Page by Treatment and<br>Biomarker | IA [1] |

# 10.7.5. Biomarker Figures

| Biomarker | Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Soluble In | flammatory Me | diators | | | |
| 2.1 | Safety | BIO_F1 | Individual Plot of Primary Soluble Inflammatory Mediators in Blood Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.2. | Safety | BIO_F1 | Individual Plot of Change from Baseline in Primary Soluble Inflammatory Mediators in Blood Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.3. | Safety | BIO_F2 | Mean (+/- SD) Plot of Primary Soluble Inflammatory Mediators in Blood Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.4. | Safety | BIO_F2 | Mean (+/- SD) Plot of Change from Baseline in Primary Soluble Inflammatory Mediators in Blood Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.5. | Safety | BIO_F1 | Individual Plot of Secondary Soluble Inflammatory Mediators in Blood Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.6. | Safety | BIO_F1 | Individual Plot of Change from Baseline in Secondary Soluble Inflammatory Mediators in Blood Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.7. | Safety | BIO_F2 | Mean (+/- SD) Plot of Secondary Soluble Inflammatory Mediators in Blood Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.8. | Safety | BIO_F2 | Mean (+/- SD) Plot of Change from Baseline in Secondary Soluble Inflammatory Mediators in Blood Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.9. | Safety | BIO_F3 | Bar Chart of Soluble Inflammatory Mediators from In-Vitro (un)stimulated Blood Pre and Post In-Vivo LPS Challenge | Generate Bar Chart Page by Treatment and Biomarker | IA [1] |
| 2.10. | Safety | BIO_F4 | Box Plot of Soluble Inflammatory Mediators from In-Vitro (un)stimulated Blood Pre and Post In-Vivo LPS Challenge | Generate Box Plot Page by Treatment and Biomarker | IA [1] |

| Biomarker | Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.11. | Safety | BIO_F1 | Individual Plot of Soluble Inflammatory Mediators in Blister Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.12. | Safety | BIO_F1 | Individual Plot of Change from Baseline in Soluble Inflammatory Mediators in Blister Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.13. | Safety | BIO_F2 | Mean (+/- SD) Plot of Soluble Inflammatory Mediators in Blister Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.14. | Safety | BIO_F2 | Mean (+/- SD) Plot of Change from Baseline in Soluble Inflammatory Mediators in Blister Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.15. | Safety | BIO_F1 | Individual Plot of Soluble Inflammatory Mediators in Urine Over Time following LPS Challenge | Page by Treatment and Biomarker | IA [1] |
| 2.16. | Safety | BIO_F1 | Individual Plot of Change from Baseline in Soluble Inflammatory Mediators in Urine Over Time following LPS Challenge | Page by Treatment and Biomarker | IA [1] |
| 2.17. | Safety | BIO_F2 | Mean (+/- SD) Plot of Soluble Inflammatory Mediators in Urine Over Time following LPS Challenge | Page by Challenge and Biomarker | IA [1] |
| 2.18. | Safety | BIO_F2 | Mean (+/- SD) Plot of Change from Baseline in Soluble Inflammatory Mediators in Urine Over Time following LPS Challenge | Page by Challenge and Biomarker | IA [1] |
| Total Leuko | cyte Numbers | 1 | | | |
| 2.19. | Safety | BIO_F1 | Individual Plot of Cell Numbers in Blood Over Time following GM-CSF Challenge | Page by Treatment and Biomarker | IA [1] |
| 2.20. | Safety | BIO_F1 | Individual Plot of Change from Baseline in Cell Numbers in Blood Over Time following GM-CSF Challenge | Page by Treatment and Biomarker | IA [1] |
| 2.21. | Safety | BIO_F2 | Mean (+/- SD) Plot of Cell Numbers in Blood Over Time following GM-CSF Challenge | Page by Challenge and Biomarker | IA [1] |

| Biomarker Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.22. | Safety | BIO_F2 | Mean (+/- SD) Plot of Change from Baseline in Cell Numbers in Blood Over Time following GM-CSF Challenge | Page by Challenge and Biomarker | IA [1] |

| Biomarker | Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Blister Volu | ıme | | | | |
| 2.23. | Safety | BIO_F5 | Bar Chart of Blister Volume Over Time | Generate Bar Chart Page by Treatment | IA [1] |
| Flow Cyton | netry | | | <u></u> | |
| 2.24. | Safety | BIO_F1 | Individual Plot of Cell Activation Markers by Flow Cytometry on Monocytes in Blood Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.25. | Safety | BIO_F1 | Individual Plot of Change from Baseline in Cell Activation Markers by Flow Cytometry on Monocytes in Blood Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.26. | Safety | BIO_F2 | Mean (+/- SD) Plot of Cell Activation Markers by Flow Cytometry on Monocytes in Blood Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.27. | Safety | BIO_F2 | Mean (+/- SD) Plot of Change from Baseline in Cell Activation Markers by Flow Cytometry on Monocytes in Blood Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.28. | Safety | BIO_F1 | Individual Plot of Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blood Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.29. | Safety | BIO_F1 | Individual Plot of Change from Baseline in Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blood Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.30. | Safety | BIO_F2 | Mean (+/- SD) Plot of Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blood Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.31. | Safety | BIO_F2 | Mean (+/- SD) Plot of Change from Baseline in Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blood Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.32. | Safety | BIO_F1 | Individual Plot of Cell Counts by Flow Cytometry in Blood Over Time | Page by Treatment and Biomarker | IA [1] |

| Biomarker | Figures | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / Example Shell | | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.33. | Safety | BIO_F1 | Individual Plot of Change from Baseline in Cell Counts by Flow Cytometry in Blood Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.34. | Safety | BIO_F2 | Mean (+/- SD) Plot of Cell Counts by Flow Cytometry in Blood<br>Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.35. | Safety | BIO_F2 | Mean (+/- SD) Plot of Change from Baseline in Cell Counts by Flow Cytometry in Blood Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.36. | Safety | BIO_F1 | Individual Plot of Cell Activation Markers by Flow Cytometry on Monocytes in Blister Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.37. | Safety | BIO_F1 | Individual Plot of Change from Baseline in Cell Activation Markers by Flow Cytometry on Monocytes in Blister Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.38. | Safety | BIO_F2 | Mean (+/- SD) Plot of Cell Activation Markers by Flow Cytometry on Monocytes in Blister Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.39. | Safety | BIO_F2 | Mean (+/- SD) Plot of Change from Baseline in Cell Activation Markers by Flow Cytometry on Monocytes in Blister Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.40. | Safety | BIO_F1 | Individual Plot of Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blister Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.41. | Safety | BIO_F1 | Individual Plot of Change from Baseline in Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blister Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.42. | Safety | BIO_F2 | Mean (+/- SD) Plot of Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blister Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.43. | Safety | BIO_F2 | Mean (+/- SD) Plot of Change from Baseline in Cell Activation<br>Markers by Flow Cytometry on Dendritic Cells in Blister Over<br>Time | Page by Challenge and Biomarker | IA [1] |

| Biomarker Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.44. | Safety | BIO_F1 | Individual Plot of Cell Counts by Flow Cytometry in Blister Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.45. | Safety | BIO_F1 | Individual Plot of Change from Baseline in Cell Counts by Flow Cytometry in Blister Over Time | Page by Treatment and Biomarker | IA [1] |
| 2.46. | Safety | BIO_F2 | Mean (+/- SD) Plot of Cell Counts by Flow Cytometry in Blister Over Time | Page by Challenge and Biomarker | IA [1] |
| 2.47 | Safety | BIO_F2 | Mean (+/- SD) Plot of Change from Baseline in Cell Counts by Flow Cytometry in Blister Over Time | Page by Challenge and Biomarker | IA [1] |

## 10.7.6. ICH Listings

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Programming Notes | Deliverable<br>[Priority] | |
| Demog | Demographic and Baseline Characteristics | | | | |
| 1. | Enrolled | DM2 | Listing of Demographic Characteristics | ICH E3 | IA [1] |

# 10.7.7. Non-ICH Listings

| Non-ICI | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Soluble | Inflammatory | Mediators | | | |
| 2. | Safety | BIO_L1 | Listing of Primary Soluble Inflammatory Mediators in Blood | | IA [1] |
| 3. | Safety | BIO_L1 | Listing of Secondary Soluble Inflammatory Mediators in Blood | | IA [1] |
| 4. | Safety | BIO_L1 | Listing of Soluble Inflammatory Mediators from In-Vitro (un)stimulated Blood | | IA [1] |
| 5. | Safety | BIO_L2 | Listing of Soluble Inflammatory Mediators in Blister | | IA [1] |
| 6. | Safety | BIO_L1 | Listing of Soluble Inflammatory Mediators in Urine following LPS Challenge | | IA [1] |
| Total Le | eukocyte Numl | pers | | | |
| 7. | Safety | BIO_L1 | Listing of Cell Numbers in Blood following GM-CSF Challenge | | IA [1] |
| Blister ' | Volume | | | | |
| 8. | Safety | BIO_L2 | Listing of Blister Volume | | IA [1] |
| Flow Cy | tometry | | | | |
| 9. | Safety | BIO_L1 | Listing of Cell Activation Markers by Flow Cytometry on Monocytes in Blood | | IA [1] |
| 10. | Safety | BIO_L1 | Listing of Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blood | | IA [1] |
| 11. | Safety | BIO_L1 | Listing of Cell Counts by Flow Cytometry in Blood | | IA [1] |
| 12. | Safety | BIO_L2 | Listing of Cell Activation Markers by Flow Cytometry on Monocytes in Blister | | IA [1] |
| 13. | Safety | BIO_L2 | Listing of Cell Activation Markers by Flow Cytometry on Dendritic Cells in Blister | | IA [1] |
| 14. | Safety | BIO_L2 | Listing of Cell Counts by Flow Cytometry in Blister | | IA [1] |

## 10.8. Appendix 8: Example Mock Shells for Data Displays

Example: BIO\_T1 Page 1 of n

Protocol: 207654 Population: Safety

Table 2.1
Summary of Primary Soluble Inflammatory Mediators in Blood

Treatment: LPS x.x ng/kg (N=xx)

Biomarker: xxxx (units)

| Visit | Planned Relative<br>Time | n | Mean | SD | Median | Min. | Max. | %CVb |
|---|---|---|---|---|---|---|---|---|
| <br>SESSION 1 DAY 1 | PRE BLISTER<br>INDUCTION | Х | X.XXX | X.XXXX | X.XXX | X.XX | X.XX | xx% |
| SESSION 1 DAY 2 | PRE FLUID<br>SAMPLING | X | x.xxx | X.XXXX | X.XXX | X.XX | X.XX | xx% |
| SESSION 1 DAY 3 | PRE FLUID<br>SAMPLING | X | X.XXX | X.XXXX | X.XXX | X.XX | X.XX | xx% |
| SESSION 2 DAY 1 | PRE BLISTER INDUCTION | х | X.XXX | X.XXXX | X.XXX | X.XX | X.XX | xx% |
| SESSION 2 DAY 1 | -5 MIN | x | X.XXX | X.XXXX | X.XXX | X.XX | X.XX | xx% |

Note: Biomarker xxxx includes <LLQ values, Biomarker yyyy includes CV>20% values, Biomarker zzzz includes Plate failed QC values (only if applicable).

Note: Values recorded as '<LLQ' have been imputed as LLQ/2 (only if applicable).

Repeat for all treatments and biomarkers

For all Summaries of Change from baseline, provide the footnote as below:

Note: Session x Day x is considered as Baseline.

Example: BIO\_F1 Protocol: 207654 Population: Safety

Figure 2.1 Individual Plot of Primary Soluble Inflammatory Mediators in Blood Over Time



S1D1=Session 1 Day 1, S1D2=Session 1 Day 2, S1D3=Session 1 Day 3, S2D1=Session 2 Day 1, S2D2=Session 2 Day 2, S2D3=Session 2 Day 3, PBI=Pre Blister Induction, PFS=Pre Fluid Sampling

Note: Biomarker xxxx includes <LLQ values, Biomarker yyyy includes CV>20% values, Biomarker zzzz includes Plate failed QC values (only if applicable).

Note: Values recorded as '<LLQ' have been imputed as LLQ/2 (only if applicable).

Repeat for all available treatments and biomarkers.

For Individual Plots of Change from baseline, provide the footnote as below:

Note: Session x Day x is considered as Baseline.

Example: BIO\_F2 Protocol: 207654 Population: Safety

Figure 2.3
Mean (+/- SD) Plot of Primary Soluble Inflammatory Mediators in Blood Over Time



S1D1=Session 1 Day 1, S1D2=Session 1 Day 2, S1D3=Session 1 Day 3, S2D1=Session 2 Day 1, S2D2=Session 2 Day 2, S2D3=Session 2 Day 3, PBI=Pre Blister Induction, PFS=Pre Fluid Sampling

Note: Biomarker xxx includes <LLQ values, Biomarker yyy includes CV>20% values, Biomarker zzzz includes Plate failed QC values (only if applicable). Note: Values recorded as '<LLQ' have been imputed as LLQ/2 (only if applicable). Repeat for all available biomarkers and challenges.

For Mean (+/- SD) Plots of Change from baseline, provide the footnote as below: Note: Session x Day x is considered as Baseline.

Example: BIO\_F3 Protocol: 207654 Population: Safety

Figure 2.9
Bar Chart of Soluble Inflammatory Mediators from In-Vitro (un)stimulated Blood Pre and Post In-Vivo LPS Challenge



Note: Biomarker xxx includes <LLQ values, Biomarker yyy includes CV>20% values, Biomarker zzzz includes Plate failed QC values (only if applicable).

Note: Values recorded as '<LLQ' have been imputed as LLQ/2 (only if applicable).

Each Bar represents a participant.

Repeat for all available treatments and biomarkers.

Example: BIO\_F4 Page 1 of n

Protocol: 207654 Population: Safety

Figure 2.10
Box Plot of Soluble Inflammatory Mediators from In-Vitro (un)stimulated Blood Pre and Post In-Vivo LPS Challenge

Treatment: x.x ng/kg (N=xx) Biomarker: xxxx(unit)



Note: Biomarker xxx includes <LLQ values, Biomarker yyy includes CV>20% values, Biomarker zzzz includes Plate failed QC values (only if applicable).

Note: Values recorded as '<LLQ' have been imputed as LLQ/2 (only if applicable).

Provide Mean, Median, Inter-quartile ranges, Minimum, Maximum and Outliers in the box plot.

Repeat for all available treatments and biomarkers.

Example: BIO\_F5
Protocol: 207654
Population: Safety

Figure 2.23
Bar Plot of Blister Volume Over Time



Note: Biomarker xxx includes <LLQ values, Biomarker yyy includes CV>20% values, Biomarker zzzz includes Plate failed QC values (only if applicable).

Note: Values recorded as '<LLQ' have been imputed as LLQ/2 (only if applicable).

Repeat for all available treatments

Example: BIO\_L1
Protocol: 207654
Population: Safety

Listing 2
Listing of Primary Soluble Inflammatory Mediators in Blood

| Treatment | Biomarker<br>(Unit) | Centre<br>ID/<br>Subj ID | Visit/<br>Planned<br>Relative<br>Time | Date/<br>Time/<br>Study<br>Day | Result | Change<br>from<br>Baseline | Test<br>Comments |
|---|---|---|---|---|---|---|---|
| LPS x.x ng/kg | xxxxxxx<br>(unit) | xxxx/<br>xxxx | xxxxx/<br>xxx<br>xxxx/<br>xxxx | xxxx/<br>xxxxx<br>xxxx/<br>xxxx | XXXX | xxxx | <llq< td=""></llq<> |
| | | | xxxx/<br>xxxx<br>xxxx/<br>xxxx | xxxx/<br>xxxx<br>xxxx/<br>xxxx | xxxx | xxxx | |
| | xxxxxx<br>(unit) | xxxx/<br>xxxx | xxxx/<br>xxxx<br>xxxx/<br>xxxx | xxxx/<br>xxxx<br>xxxx/<br>xxxx | xxxx | xxxx | CV>20%<br>>ULQ |

Note: LLQ=Lower Limit of Quantification, ULQ=Upper Limit of Quantification, CV=Coefficient of Variation.

Note: Repeat for all available treatments and biomarkers.

207654 Example: BIO\_L2 Page 1 of n

Protocol: 207654 Population: Safety

Listing 5

| Listing of Soluble Inflammatory Mediators in Blister | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment | Biomarker<br>(Unit) | Centre<br>ID/<br>Subj<br>ID | Visit/<br>Planned<br>Relative<br>Time | Date/<br>Time/<br>Study<br>Day | Årm | Result | | Test<br>Comments |
| LPS x.x<br>ng/kg | xxxxxx<br>(unit) | xxxx/<br>xxxx | xxxxx/<br>xxx | xxxx/<br>xxxx/<br>xxxxx | Right | XXXX | | <llq< td=""></llq<> |
| | | | | xxxx/<br>xxxx/<br>xxxxx | Left | XXXX | | |
| | | | | xxxx/<br>/xxxxx | Average | XXXX | XXXX | |
| | | | xxxx/<br>xxxx | xxxx/<br>xxxx/<br>xxxx | Right | XXXX | XXXX | >ULQ |
| | | | | xxxx/<br>xxxx/<br>xxxx | Left | XXXX | | |
| | | | | xxxx/<br>/xxxxx | Average | XXXX | XXXX | |

Note: LLQ=Lower Limit of Quantification, ULQ=Upper Limit of Quantification, CV=Coefficient of Variation.

Note: Repeat for all available treatments and biomarkers.